CLINICAL TRIAL: NCT01449968
Title: Provision of a Mobile Geriatric Team Extra-Community Hospital in Assessing and Regulating the Hospitalization of Frail Elderly Patients With Complex Medical and Social Situation
Brief Title: Provision of a Mobile Geriatric Team Extra-Community Hospital
Acronym: UMG
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurCIC, Pr Pascal COUTURIER, University Hospital, Grenoble, University Hospital, Grenoble
Other Study IDs: DCIC 10 16
Record Dates: First submitted 2011-07-07; First posted 2011-10-10 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Geriatric Disorder; Mobil Unit
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- home visit of UMG: home visit with evaluation and management of the situation (control over in-home telephone)
  Interventions: Other: home visit
- telephone management: geriatric mobile unit provides a telephone advice only to the general practitioner with guidance and recommendations (call control)
  Interventions: Other: telephone management

INTERVENTIONS:
Other: home visit — home visit of UMG
  Groups: home visit of UMG
Other: telephone management — telephone management of the situation reported by the patient's GP
  Other Names: telephone management of the mobile unit of Geriatrics
  Groups: telephone management

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of the mobile unit to reduce the geriatric hospital inappropriate (especially for emergencies) to 1 month.

The primary endpoint: survival without hospitalization through the emergency inappropriate to 1 month.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of the Mobile Geriatrics on the management of complex situations in retirement homes and in ambulatory care of frail elderly patients, reported by the generalist doctor, in terms of improving the conditions of use technical support hospital follow-up recommendations given by the mobile team and their impact on outcomes of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 and over living in complex medical or psycho-social complex or at risk of hospitalization
* Patient affiliated to social security or beneficiary of such a regime
* Patient available for follow-up to 6 months with a caregiver or accompanying social duly appointed.

Exclusion Criteria:

* Patient residing outside intervention sector
* Life-threatening emergency (ambulance)
* Lack of complexity of the situation, supported by routine care

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes patients over 75 years in medical condition or psycho-social complex, followed by a general practitioner to population centers include: Grenoble, Annecy and Roanne.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
effectiveness of the visit of the mobile unit to reduce the geriatric hospital inappropriate (especially for emergencies) to 1 month | 1 month
  inappropriate survival without hospitalization through the emergency room at 1 month

SECONDARY OUTCOMES:
follow-up rate of the proposals of UMG ext (adherence to recommendations and feasibility) and analyze the reasons for not monitoring these proposals one month | 1 month
  follow-up of recommendations made by the mobile unit of Geriatrics
survival without hospitalization inappropriate, mortality, changes in functional status and cognitive health care consumption up to 6 months of surgery | 6 months
  Unplanned hospitalization rates obtained by telephone follow-up at 3 and 6 months
effectiveness of the visit of the mobile geriatric home versus telephone follow-up of mobile geriatric unit | 6 months
  Analysis of sub-groups
needs and difficulties of attending physicians in the care of frail elderly patients with complex medical and social situation before and after the establishment of mobile units for geriatrics. | 1 year
  Questionnaire to GPs in the health sector concerned
cost effectiveness of two types of visit of the mobile unit of Geriatrics (telephone regulation and control over travel home phone) | 6 months
  Cost of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal COUTURIER, PUPH, Principal Investigator — Geriatric unit - University Hospital of Grenoble
Locations (3):
- France (3):
  - CH Annecy, Annecy
  - University Hospital of Grenoble, Grenoble
  - CH Roanne, Roanne

REFERENCES:
- [Background] Bernabei R, Landi F, Gambassi G, Sgadari A, Zuccala G, Mor V, Rubenstein LZ, Carbonin P. Randomised trial of impact of model of integrated care and case management for older people living in the community. BMJ. 1998 May 2;316(7141):1348-51. doi: 10.1136/bmj.316.7141.1348. PMID 9563983
- [Background] Stuck AE, Siu AL, Wieland GD, Adams J, Rubenstein LZ. Comprehensive geriatric assessment: a meta-analysis of controlled trials. Lancet. 1993 Oct 23;342(8878):1032-6. doi: 10.1016/0140-6736(93)92884-v. PMID 8105269
- [Background] Elkan R, Kendrick D, Dewey M, Hewitt M, Robinson J, Blair M, Williams D, Brummell K. Effectiveness of home based support for older people: systematic review and meta-analysis. BMJ. 2001 Sep 29;323(7315):719-25. doi: 10.1136/bmj.323.7315.719. PMID 11576978